CLINICAL TRIAL: NCT04120519
Title: Thalidomide, Cyclophosphamide and Dexamethasone for Adult Patients With Recurrent/Refractory Langerhans Cell Histiocytosis: A Single Arm, Single Center, Prospective Phase 2 Study
Brief Title: Thalidomide, Cyclophosphamide and Dexamethasone for Recurrent/Refractory Adult Langerhans Cell Histiocytosis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Cao Xinxin, Associate Professor, Peking Union Medical College Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PUMCHRRLCH-1
Record Dates: First submitted 2019-10-07; First posted 2019-10-09 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-06

CONDITIONS: Langerhans Cell Histiocytosis
Keywords: Langerhans cell histiocytosis; adult; recurrent/refractory
MeSH Terms: conditions — Histiocytosis, Langerhans-Cell; Recurrence | interventions — Dexamethasone; Cyclophosphamide

STUDY DESIGN:
Intervention Model Description: thalidomide combined with dexamethasone and cyclophosphamide
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TCD (Experimental): thalidomide 100mg qn cyclophosphamide 300mg/m2 d1,8,15 dexamethasone 40mg d1,8,15,22
  Interventions: Drug: thalidomide combined with dexamethasone and cyclophosphamide

INTERVENTIONS:
Drug: thalidomide combined with dexamethasone and cyclophosphamide — TCD

SUMMARY:
Langerhans cell histiocytosis (LCH) is a rare, heterogeneous histiocytic disorder occurring most commonly in children. Because of the rarity of LCH in adults and a lack of prospective randomized trials, the treatment strategy for adults is mostly based on pediatric protocols. The overall response rate of therapy based on vinblastine plus prednisone in adults is lower than in children and the treatment tends to show higher toxicity.There is little data to guide therapy after frontline treatment. In a phase 2 trial, thalidomide as monotherapy gave a 70% response rate in recurrent/refractory low risk LCH but there were no responses in six high risk children. We want to analyze the efficacy and toxicity of thalidomide combined with dexamethasone and cyclophosphamide regimens in the treatment of recurrent/refractory LCH among adult patients at our hospital.

ELIGIBILITY:
Inclusion Criteria:

* • Histologically confirmed diagnosis of LCH.

  * Patients were recurrent/refractory or at least receive one line of systemic treatment of LCH
  * Age ≥18 years and ≤75 years.
  * LCH involved multisystem or multifocal single system.
  * Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
  * Patients must have adequate renal, liver, and bone marrow function as defined by the following criteria:

    * Absolute neutrophil count ≥1500 cells per mm3 or ≥500 cells per mm3 in the case of known hematopoietic system involvement by LCH.
    * Platelet count ≥100000 cells per mm3 or ≥20000 cells per mm3 in the case of known hematopoietic system involvement by LCH.
    * Creatinine clearance [according to Cockcroft formula] ≥60 mL/min.
    * Aspartate aminotransferase and alanine aminotransferase ≤2·5×upper limit of normal [ULN], and total bilirubin ≤2·5×ULN; or ≤10×ULN in the case of known liver involvement by LCH.
  * No active or untreated infection.
  * No cardiac abnormalities.
  * Subject provide written informed consent.
  * A female is eligible to enter and participate in this study if she is of:

    * Non-childbearing potential including ω Any female who has had a surgical procedure rendering her incapable of becoming pregnant.

ω Subjects have experienced total cessation of menses for more than 1 year and be greater than 45 years in age.

⎫ Childbearing potential, including any female who has had a negative serum pregnancy test within 2 weeks prior to the first dose of study treatment, and agrees to use adequate contraception.

• Male subjects must use an effective barrier method of contraception during the study and for 90 days following the last course of MA if sexually active with a childbearing potential

Exclusion Criteria:

* • Non-langerhans cell histiocytosis.

  * Patients had concurrent malignancies.
  * Patients who were newly diagnosed LCH.
  * History of myocardial infarction, or unstable angina, or New York Heart Association (NYHA) Grade III-IV within 6 months prior to Day 1.
  * Women who were pregnant or of childbearing potential.
  * Known HIV seropositive, active hepatitis C infection, and/or hepatitis B (defined as HCV RNA

    ≥103 copies or HBV DNA ≥103 copies at screening).
  * Major surgical procedure within 28 days prior to the first dose of study treatment.
  * Presence of uncontrolled infection.
  * Evidence of active bleeding or bleeding diathesis.
  * Any serious and/or unstable pre-existing medical, psychiatric, or other condition that could interfere with subject's safety, provision of informed consent, or compliance to study procedures.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-10-10 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Event-free survival | the duration from initiation of treatment to the date of first documented event or date of death from any cause, whichever come first, assessed up to 5 years
  Events were defined as a poor response to TCD, reactivation after TCD therapy and death from any cause.

SECONDARY OUTCOMES:
Overall response rate | on 12 months
  the cumulative number of patients with either non-active disease or regressive disease (signs and symptoms were improved with no new lesions) after TCD therapy
Overall survival | the duration from initiation of TCD treatment to the date of death or last follow-up, assessed up to 5 years
  Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Jian Li, Study Director — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, China